CLINICAL TRIAL: NCT05048303
Title: Multicenter Clinical Cohort Study of Modified Flexible Fixation Latarjet Procedure for Recurrent Shoulder Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUWEI
Record Dates: First submitted 2021-07-27; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Dislocation
Keywords: shoulder dislocation; Latarjet procedure; graft remodeling
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: A multi-center, prospective, single-arm clinical intervention cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized Lutajet operative group (Experimental): Arthroscopic modified individualized flexible Latarjet procedure with preservation of the coracoacromial arch. During the procedure, we perform coracoid osteotomy with preservation of coracoacromial arch, then split subscapular tendon, transfer the bone graft and fix it with double button under arthroscopy.
  Interventions: Procedure: Arthroscopic modified individualized flexible Latarjet procedure

INTERVENTIONS:
Procedure: Arthroscopic modified individualized flexible Latarjet procedure — The modifications were as follows: (1)the coracoid graft and conjoint tendon were prepared using a mini-open technique with an incision of 2.5 cm and coracoacromial ligament were preserved. A total of 2 bone tunnels were drilled. (2)The anterior (including part of the incision used for obtaining the graft), standard antelateral, and posterior portals were set. (3) The glenoid was marked at the 4-o'clock position, and then the subscapularis muscle was split. (4)The glenoid tunnel was drilled where the suture linked to the graft was passed, and the graft was pulled to the glenohumeral joint via the sutures. A knotless suture anchor for antirotation (PushLock; Arthrex) was fixed to the glenoid to prevent rotation of the graft.

SUMMARY:
The shoulder joint is the most flexible joint of human body and shoulder joint dislocation is the most common joint dislocation of human body. Currently, there are different treatments for anterior shoulder dislocation, but for young patients with high sports requirements and apparent glenoid defect, soft tissue repair is not enough otherwise patients will suffer a high recurrent rate.

In 1954, M. Latarjet invented the coracoid process osteotomy and transposition technique, called the Latarjet procedure, which was a bony repair technique and was later promoted by G. Walch. This technique not only reconstructs the defect glenoid, the sling effect attached to the conjoint tendon also strengthens the anterior and inferior structure. Due to the advantages of low recurrence rate after Latarjet procedure, high rate of patients returning to sports and high satisfaction, it has become the only surgery that has been widely used in more than ten similar surgeries in history. In 2007, French physician Lafosse successfully completed the technique under arthroscopy. However, this surgery traditionally uses screws to fix the bone block, but screw fixation has difficulties like exposed nail head, uncertain bone block positioning, and high absorption rate of the bone block. In 2012, P.Boileau further improved this technique, innovating to avoid the above-mentioned complications through suture button fixation. However, since the Latarjet procedure was invented for decades, scholars have been worried about the unavoidable defects of this technique including the destruction of the coracoacomial arch, pectoralis minor injury and a series of complications caused by non-anatomical reconstruction of the glenoid.

In order to further develop this technology, make it more simple, easy to promote, and safer, based on our clinical and basic research on flexible fixation Latarjet technique for more than 8 years, we have innovatively developed an individualized and improved flexible fixation Latarjet technique that preserves the coracoacomial arch. We assumed that our modified technique, which retains the coracoacomial arch, 1) has the same satisfactory clinical effect. 2) The individualized reconstruction of glenoid defect is more identical with the biomechanics of the shoulder joint. The bone block will finally be remodeled according to the best fit circle. 3) The tiny subscapular tendon split is less damaged and safer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-59 years, gender unlimited.
* Patients with recurrent shoulder dislocation who were judged by clinicians to be suitable for modified flexible fixation Latarjet procedure according to surgical indications (1. Glenoid bone defect>20% 2. Glenoid defect>15% and ISIS>6 3. Glenoid defect>10% and competitive athletes)
* Volunteers to join the study and sign informed consent

Exclusion Criteria:

* Clinical and imaging diagnosis combined with other shoulder diseases, such as frozen shoulder, rotator cuff injury, shoulder joint degeneration.
* Basic diseases of important organs ( including severe osteoporosis, dysfunction of important organs, connective tissue diseases, neuropsychiatric disorders, epilepsy, etc. )

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 364 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Rowe Score | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  Dr. Carter R. Rowe, an orthopedic shoulder specialist at the Massachusetts General Hospital in Boston, USA, proposed in the JBJS magazine in the United States in 1978 that the Rowe score scale for the evaluation of the clinical effects of repair surgery for shoulder joint instability. Including stability, mobility and functional evaluation, the higher the score, the higher the stability and the better the shoulder function.

SECONDARY OUTCOMES:
Change in the ASES score | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  The ASES (American Association of Shoulder and Elbow Surgery scores) are the shoulder joint function evaluation standards adopted by the American Association of Shoulder and Elbow Surgeons in 1993. The system is a percentile system that needs to be converted. The pain in the assessment part of the patient and the cumulative daily activities each account for 50%. The full score is 100 points. The higher the score, the better the shoulder joint function.
Change in the Constant-Murley score | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  The Constant-Murley Shoulder Scoring Scale was designed by Christopher Constant and Alan Murley in 1986. It is mainly used to assess the severity of shoulder-related diseases. The scale has good reliability and validity, including pain and function. , Mobility and muscle strength, the total score is 100, the higher the score, the better the function.
Change in the Visual Analogue Scale | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  The visual analogue scale (VAS) is used for pain assessment. It is widely used in clinical practice in China. The basic method is to use a moving ruler about 10cm long, with 10 scales on one side, and the two ends are respectively "0" and "10" points. A point of 0 means no pain. A score of 10 represents the most severe pain that is unbearable.
Change in the Range of Motion | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  The degree of movement of the shoulder joint can reflect the recovery of shoulder joint function, including flexion, extension, abduction, adduction, external rotation and internal rotation.
Change in the bone healing | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  Through CT scan and 3D reconstruction, we detect the change of bone healing and reshaping during different time period.
Change in the Samilson-Prieto score | Preoperative, Day 1, Month 6, Month 12, Month 18, Month 24
  Through X ray of true AP view to evaluate the degeneration of the shoulder joint

IPD SHARING:
Plan to Share IPD: No